CLINICAL TRIAL: NCT02409693
Title: Retrospective Analysis of Perioperative Anesthetic Care and Analgesia Management of Patient Undergoing Bilateral Myringotomy With Tube Insertion
Status: Withdrawn | Type: Observational
Why Stopped: Unable to obtain funding
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Richard Cartabuke, Co-Director Outpatient Anesthesia Services, Nationwide Children's Hospital
Other Study IDs: IRB15-00179
Record Dates: First submitted 2015-03-30; First posted 2015-04-07 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Otitis Media With Effusion (OME)
MeSH Terms: conditions — Otitis Media with Effusion | interventions — Middle Ear Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Myringotomy with tube insertion: Patients who received surgically inserted ear tubes.
  Interventions: Procedure: Myringotomy with tube insertion

INTERVENTIONS:
Procedure: Myringotomy with tube insertion
  Other Names: BTI

SUMMARY:
This is a retrospective chart review. The purpose of this study is to retrospectively examine the use of perioperative analgesics on the incidence of postoperative pain and emergence delirium in patients undergoing bilateral myringotomy with tube insertion (BTI), as well as events associated with treatment including postoperative vomiting and time to discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent myringotomy with tube insertion from January 1, 2015 through February 28, 2015 at NCH.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have undergone anesthesia for surgical ear tube placement at Nationwide Children's Hospital from January 1, 2015 through February 28, 2015.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain scores | 1 hr post-op
  Wong-Baker FACES and/or the Face, Legs, Activity, Cry, Consolability (FLACC) pain scores

SECONDARY OUTCOMES:
Presence of emergence delirium | 1 hr post-op
  Agitation when awakening from anesthesia
Post-operative nausea & vomiting | 1 hr post-op
  Incidence of nausea and vomiting in the post-anesthesia care unit (PACU)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Cartabuke, MD, Principal Investigator — Nationwide Children's Hospital